CLINICAL TRIAL: NCT05886153
Title: Verification Protocol for the Cloud DX Vitaliti Continuous Vital Signs Monitor (Model CVSM-1A) for Clinical Use and Self Measurement in Ambulatory Settings
Brief Title: Verification Protocol for the Cloud DX Vitaliti Continuous Vital Signs Monitor (VERDICT-2)
Acronym: VERDICT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); Population Health Research Institute (Other); Cloud DX Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: v2.0_2023-01-05
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Blood Pressure; Respiration; Pulse Rate; Oxygen Saturation; Temperature; Heart Rate
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Single group verification testing of the Vitaliti Continuous Vital Sign Monitor Model CVSM-1A device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitaliti CVSM Device (Other): Examine the accuracy of the Cloud DX Vitaliti Continuous Vital Signs Monitor (Model: CVSM-1A) in an ambulatory context with healthy participants to determine the accuracy of continuous non-invasive vital signs metrics including respiration, pulse rate, oxyhemoglobin saturation (SpO2), core temperature, heart rate, and cNIBP against standard comparator devices guided by consensus standards.
  Interventions: Device: Vitaliti Continuous Vital Sign Monitor Model CVSM-1A

INTERVENTIONS:
Device: Vitaliti Continuous Vital Sign Monitor Model CVSM-1A — Measurements recorded by the Vitaliti CVSM device will be compared to the recordings from various standardized comparator devices.

SUMMARY:
The VERDICT-2 verification study will examine the accuracy of the Cloud DX Vitaliti Continuous Vital Signs Monitor (Model: CVSM-1A) in an ambulatory context with healthy participants. The objective is to determine the accuracy of continuous non-invasive vital signs metrics including respiration, pulse rate, oxyhemoglobin saturation (SpO2), core temperature, heart rate, and cNIBP against standard comparator devices guided by consensus standards.

DETAILED DESCRIPTION:
Effective postoperative care is faced with several challenges- patients experience major complications following surgery, which often require re-hospitalization or utilization of healthcare services (i.e., emergency room visits) once discharged into the community. New remote automated monitoring (RAM) technologies that enable data integration, synthesis, and real-time alerts to clinicians have the potential to transform postoperative care, similar to how intraoperative care has evolved.

The Cloud DX Vitaliti Continuous Vital Signs Monitor (Model: CVSM-1A) is a continuous vital sign monitor intended to measure vital metrics including systolic and diastolic blood pressures (via ECG/ photoplethysmography [PPG]), pulse (via PPG), respiration rate (via impedance respiration waveform), core body temperature (via infrared sensor), and blood oxygen saturation levels (via PPG) of an adult individual using non-invasive techniques.

The VERDICT-2 verification study will examine the accuracy of the Vitaliti CVSM in an ambulatory context with healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Healthy participant (no known significant health problems)
3. Provide informed consent to participate

Exclusion Criteria:

1. Active smoker
2. Recent exposure to carbon monoxide
3. Have unexplained shortness of breath at rest
4. Pregnant
5. Hearing aid/Cochlear Implant
6. Current arrhythmia
7. ICD/Pacemaker
8. Current respiratory disease/infection
9. Significant body tremors/shaking
10. Epilepsy
11. History of unexplained fainting/syncope
12. Have any disorder that prohibits placement of the device (i.e., skin rash/abrasion, open or infected sore)
13. Cerebrospinal Fluid Shunt
14. Unable to ambulate, stand, or lay in supine position
15. Allergy to adhesive
16. Unable to understand or speak English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Respiration Rate | 44 Minutes
  Determining the accuracy of the impedance respiration waveform on the Vitaliti device to measure respiration rate, compared to an appropriate standardized comparator device. The Vitaliti CVSM will be evaluated against performance criteria determined to be clinically relevant, in alignment with predicate devices, and as defined by the manufacturer, since there are no internationally recognized consensus standards.
Pulse Rate | 27 Minutes
  Determining the accuracy of the ECG/photoplethysmography (PPG) on the Vitaliti device to measure pulse rate, compared to an appropriate standardized comparator device. Detailed analysis will be conducted to verify accuracy of the Vitaliti device against performance criteria as defined in IEC 60601-2-27:2011/ (R2016).
Oxyhemoglobin Saturation | 27 Minutes
  Determining the accuracy of the electrocardiogram (ECG)/photoplethysmography (PPG) on the Vitaliti device to measure blood oxygen saturation, compared to an appropriate standardized comparator device. A detailed analysis will be performed to compare the Vitaliti device against performance criteria as defined in ISO 80601-2-61:2017, MOD.
Temperature | 12 Minutes
  Determining the accuracy of the infrared sensor on the Vitaliti device to measure core body temperature, compared to an appropriate standardized comparator device. A detailed analysis will be conducted to verify accuracy of the Vitaliti device against performance criteria as defined in ISO 80601-2-56:2017/AMD-1:2018.
Heart Rate | 36 Minutes
  Determining the accuracy of the electrocardiogram (ECG) on the Vitaliti device to measure heart rate, compared to an appropriate standardized comparator device. A detailed analysis will be conducted to verify accuracy of the Vitaliti device against performance criteria as defined in IEC 60601-2-27:2011/ (R2016).
Blood Pressure | 30 Minutes
  Determining the accuracy of the electrocardiogram (ECG)/photoplethysmography (PPG) on the Vitaliti device to measure blood pressure, compared to an appropriate standardized comparator device. A detailed analysis will be conducted to verify accuracy against performance criteria as defined in ISO 81060-2: 2018/AMD-1:2020.

CONTACTS AND LOCATIONS:
Overall Officials: Maura Marcucci, M.D., MSc, Principal Investigator — McMaster University, Population Health Research Institute; Michael McGillion, PhD, Principal Investigator — McMaster University, Population Health Research Institute
Locations (1):
- McMaster University, Hamilton, Ontario, Canada